CLINICAL TRIAL: NCT03212326
Title: Contrast Enhanced Intracardiac Echocardiography (ICE) for Localization of Myocardial Scar During Ablation of Ventricular Tachycardia
Brief Title: Contrast ICE for Myocardial Scar in VT Ablations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1205012398
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definity (Experimental): Perflutren echo contrast is infused to enhance intracardiac echo imaging recorded during catheter ablation of ventricular tachycardia. We will compare areas that appear to be myocardial scar on ultrasound with areas of abnormal electrical signals obtained by direct catheter mapping.
  Interventions: Drug: Perflutren Lipid Microsphere Intravenous Suspension [DEFINITY]

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere Intravenous Suspension [DEFINITY] — Perflutren 1.3mL diluted in 50 mL is infused intravenously, and intracardiac echo imaging is recorded to analyze for areas of possible myocardial scar, which is then compared with areas of abnormal electrical signal via direct catheter mapping which is performed during ablation of ventricular tachycardia.

SUMMARY:
There is a high correlation between scar areas identified by contrast-enhanced ICE and scar areas identified by conventional electroanatomic mapping. Therefore, the investigators will assess the utility of contrast-enhanced ICE to identify and localize myocardial scar real-time during VT ablation procedures.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a life-threatening arrhythmia which occurs frequently in the setting of structural heart disease, most often as result of myocardial fibrosis or scar. Catheter ablation is often performed to treat recurrent VT, but is predicated on precise localization of myocardial scar, as scar is often the source of VT. Currently during VT ablation procedures the identification of scar is based on electroanatomic mapping where bipolar voltage criteria have been established (i.e., bipolar electrogram voltage < 1.5 mV is considered scar). However this definition is purely based on electrical signal information and so has significant limitations: 1) there has not been definitive establishment of the sensitivity and specificity of this threshold for defining scar in comparison with tissue; 2) a detailed 3-D map created by time-consuming movement of the mapping catheter must be obtained in order to assess the existence and location of the scar; 3) only scar on the surface in contact with the mapping catheter (most often endocardial) may be definitively identified, whereas there may be intramyocardial or epicardial scar that would not be identified unless the mapping catheter makes direct contact with those areas which may involve additional risky access (epicardial) or even impossible (intramyocardial). For these reasons it would be very helpful to have another method to identify and localize myocardial scar during a VT ablation procedure. Cardiac MRI has been validated for identifying and localizing scar, but would not be recommended for many patients due to presence of ICD (implantable cardioverter-defibrillator) devices in these patients. Contrast-enhanced echocardiography has been validated to identify myocardial scar (Montant 2010), and intracardiac echocardiography (ICE) is standardly used in VT ablation procedures. Therefore, the investigators will assess the utility of contrast enhanced ICE by identifying and localizing myocardial scar real-time during VT ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject is undergoing catheter ablation of likely reentrant VT
* Planned use of intracardiac echocardiography (ICE)
* Subject is willing to sign and date the study informed consent form

Exclusion Criteria:

* Contraindication to Perflutren (Optison) echo contrast
* Known right-to-left, bidirectional, or transient right-to-left cardiac shunts
* Known hypersensitivity to Perflutren, blood, blood products or albumin
* Subject has medical condition that would limit study participation (as per MD discretion)
* Subject is pregnant
* Inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Liu, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from hospital inpatient ward and from electrophysiology laboratory procedure suites. Recruitment commenced March 2013, and ended March 2016.
Period: Overall Study
Arm/Group | Definity
Started | 24
Completed | 20
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Definity
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24
left ventricular ejection fraction among subjects [Median (Inter-Quartile Range); unit: percent] | 25 [20 to 31.5]
number of subjects with hypertension [Count of Participants; unit: Participants] | 10
number of subjects with implanted defibrillator [Count of Participants; unit: Participants] | 21
number of subjects with ischemic cardiomyopathy [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Myocardial Scar on Echo and Voltage Maps
Description: location of left ventricular myocardial scar and abnormal electrograms
Time Frame: day 0 (intraoperative: data collected during the mapping procedure)
Population: 3 of 24 enrolled subjects did not have voltage mapping, and 1 of 24 subjects did not have echo contrast injection; thus a total of 4 subjects did not have both echo contrast and voltage mapping in order to allow scar comparison; therefore the 20 subjects with complete echo and voltage maps were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Definity
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Number of Subjects With Ventricular Tachycardia Mapped
Description: If ventricular tachycardia was induced and mapped then this counts as yes
Time Frame: day 0 (intraoperative: data collected during the mapping procedure)
Population: 4 of 24 enrolled subjects did not inducible ventricular tachycardia; thus a total of 4 subjects did not have both scar and ventricular tachycardia mapping in order to allow scar comparison; therefore the 20 subjects with complete scar and ventricular tachycardia maps were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Definity
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Definity
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03212326/Prot_SAP_000.pdf